CLINICAL TRIAL: NCT01140061
Title: A 3-Part Study to Evaluate Safety, Tolerability, and Pharmacokinetics of MK-0873 Following Cumulative Patch and Repeated Max Area Applications in Healthy Subjects and Psoriasis Patients
Brief Title: Safety, Tolerability and Pharmacokinetics of MK-0873 Following Patch Application in Healthy Participants and Psoriasis Participants (MK-0873-020)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0873-020
Record Dates: First submitted 2010-06-07; First posted 2010-06-09 (Estimated); Results first posted 2014-12-12 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2019-01

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (10):
- Panel A - MK-0873 5.1 mg (Experimental): In Part I, healthy participants received skin patches containing nothing (plain patch), placebo, and various potencies of MK-0873 cream (0.05%, 0.5%, or 2%; yielding a dose of 5.1 mg of MK- 0873) once daily for 21 days.
  Interventions: Drug: MK-0873 Patch; Drug: Placebo Patch; Drug: Plain patch
- Panel A - Placebo (Placebo Comparator): In Part I, healthy participants received skin patches containing nothing (plain patch) or placebo once daily for 10 days.
  Interventions: Drug: Placebo Patch; Drug: Plain patch
- Panel B - MK-0873 25 mg (Experimental): In Part II, healthy participants received skin application of 0.5% MK-0873 cream (yielding a dose of 25 mg of MK- 0873) twice daily for 10 days.
  Interventions: Drug: MK-0873 Cream
- Panel B - Placebo (Placebo Comparator): In Part II, healthy participants received skin application of placebo cream twice daily for 10 days.
  Interventions: Drug: Placebo Cream
- Panel C - MK-0873 100 mg (Experimental): In Part II, healthy participants received skin application of 2% MK-0873 cream (yielding a dose of 100 mg of MK-0873) once daily for 10 days.
  Interventions: Drug: MK-0873 Cream
- Panel C - Placebo (Placebo Comparator): In Part II, healthy participants received skin application of placebo cream once daily for 10 days.
  Interventions: Drug: Placebo Cream
- Panel D - MK-0873 200 mg (Experimental): In Part II, healthy participants received skin application of 2% MK-0873 (yielding a dose of 100 mg of MK-0873) twice daily for 10 days.
  Interventions: Drug: MK-0873 Cream
- Panel D - Placebo (Placebo Comparator): In Part II, healthy participants received skin application of placebo cream twice daily for 10 days.
  Interventions: Drug: Placebo Cream
- Panel E and Extension - MK-0873 200 mg (Experimental): In Part III, participants with mild psoriasis received skin application of 2% MK-0873 cream (yielding a dose of 100 mg of MK-0873) twice daily for up to 28 days.
  Interventions: Drug: MK-0873 Cream
- Panel E and Extension - Placebo (Placebo Comparator): In Part III, participants with mild psoriasis received skin application of placebo cream twice daily for up to 28 days.
  Interventions: Drug: Placebo Cream

INTERVENTIONS:
Drug: MK-0873 Patch — MK-0873 skin patches containing 0.05%. 0.5%, or 2% MK-0873
  Arms: Panel A - MK-0873 5.1 mg
Drug: MK-0873 Cream — MK-0873 cream containing 0.05%, 0.5%, or 2% MK-0873
  Arms: Panel B - MK-0873 25 mg; Panel C - MK-0873 100 mg; Panel D - MK-0873 200 mg; Panel E and Extension - MK-0873 200 mg
Drug: Placebo Patch — Placebo patches matching MK-0873 0.05%, 0.5%, or 2% patches
  Arms: Panel A - MK-0873 5.1 mg; Panel A - Placebo
Drug: Placebo Cream — Placebo cream matching MK-0873 0.05%, 0.5%, or 2%
  Arms: Panel B - Placebo; Panel C - Placebo; Panel D - Placebo; Panel E and Extension - Placebo
Drug: Plain patch — Plain patch containing no MK-0873 or placebo
  Arms: Panel A - MK-0873 5.1 mg; Panel A - Placebo

SUMMARY:
This study will evaluate the incidence of erythema and other local cutaneous irritation after administration of MK-0873 by patch or cream formulation in healthy participants and participants with mild psoriasis. Part I and Part II in healthy participants will be initiated prior to Part III in psoriasis participants. The primary hypotheses of the study are: 1) that MK-0873 is safe and well tolerated in healthy participants and participants with psoriasis and 2) that the maximum plasma concentration of MK-0873 is <20 nM in healthy participants and participants with psoriasis.

ELIGIBILITY:
Inclusion Criteria:

Part I, II and III:

* Female participants of reproductive potential must test negative for pregnancy and agree to use two acceptable methods of birth control;
* In good general health;
* Nonsmoker;

Part III only:

* Has diagnosis of plaque-type psoriasis, and has lesions covering at least 3% of total body surface area;

Exclusion Criteria:

Part I, II and III:

* Has a history of stroke, chronic seizures or major neurological disease;
* Has a history of cancer;
* Is a nursing mother;

Part III only:

* Has nonplaque forms of psoriasis;
* Has current drug-induced psoriasis;
* Has received phototherapy, systemic medications/treatments, or used topical medication that could affect psoriasis;
* Has used any systemic immunosuppressants or biologics within the past 4 weeks.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2010-05-01 (Actual); Primary Completion 2011-03-01 (Actual); Study Completion 2011-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=0873-020&kw=0873-020&tab=access

RESULTS

PARTICIPANT FLOW:
Groups:
- Panel A - MK-0873 5.1 mg: In Part I, healthy participants received skin patches containing nothing (plain patches), placebo, and various potencies of MK-0873 cream (0.05%, 0.5%, or 2%; yielding a dose of 5.1 mg MK-0873) once daily for 21 days.
- Panel A - Placebo: In Part I, healthy participants received skin patches containing nothing (plain patch) and placebo once daily for 21 days.
- Panel B - MK-0873 25 mg: In Part II, healthy participants received skin application of 0.5% MK-0873 cream (yielding a dose of 25 mg of MK-0873) twice daily for 10 days.
Period: Part I
Arm/Group | Panel A - MK-0873 5.1 mg | Panel A - Placebo | Panel B - MK-0873 25 mg | Panel B - Placebo | Panel C - MK-0873 100 mg | Panel C - Placebo | Panel D - MK-0873 200 mg | Panel D - Placebo | Panel E and Extension - MK-0873 200 mg | Panel E and Extension - Placebo
Started | 7 (Includes 1 replacement participant) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 6 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part II
Arm/Group | Panel A - MK-0873 5.1 mg | Panel A - Placebo | Panel B - MK-0873 25 mg | Panel B - Placebo | Panel C - MK-0873 100 mg | Panel C - Placebo | Panel D - MK-0873 200 mg | Panel D - Placebo | Panel E and Extension - MK-0873 200 mg | Panel E and Extension - Placebo
Started | 0 | 0 | 6 | 2 | 6 | 2 | 6 | 2 | 0 | 0
Completed | 0 | 0 | 6 | 2 | 6 | 2 | 6 | 2 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part III
Arm/Group | Panel A - MK-0873 5.1 mg | Panel A - Placebo | Panel B - MK-0873 25 mg | Panel B - Placebo | Panel C - MK-0873 100 mg | Panel C - Placebo | Panel D - MK-0873 200 mg | Panel D - Placebo | Panel E and Extension - MK-0873 200 mg | Panel E and Extension - Placebo
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 2 (Includes 1 replacement participant)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Extension
Arm/Group | Panel A - MK-0873 5.1 mg | Panel A - Placebo | Panel B - MK-0873 25 mg | Panel B - Placebo | Panel C - MK-0873 100 mg | Panel C - Placebo | Panel D - MK-0873 200 mg | Panel D - Placebo | Panel E and Extension - MK-0873 200 mg | Panel E and Extension - Placebo
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 2
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Laboratory Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Panel A - MK-0873 5.1 mg | Panel A - Placebo | Panel B - MK-0873 25 mg | Panel B - Placebo | Panel C - MK-0873 100 mg | Panel C - Placebo | Panel D - MK-0873 200 mg | Panel D - Placebo | Panel E and Extension - MK-0873 200 mg | Panel E and Extension - Placebo | Total
Number analyzed (Participants) | 7 | 2 | 6 | 2 | 6 | 2 | 6 | 2 | 7 | 2 | 42
Age, Continuous [Mean (Full Range); unit: Years] | 42.71 (12.19) [23 to 53] | 30.50 (17.68) [18 to 43] | 40.00 (11.78) [26 to 60] | 45.50 (14.85) [35 to 56] | 45.67 (12.79) [28 to 62] | 34.00 (7.07) [29 to 39] | 30.33 (6.77) [21 to 38] | 35.50 (2.12) [34 to 37] | 42.86 (11.33) [23 to 54] | 40.00 (15.56) [29 to 51] | 39.67 (11.49) [18 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 3 | 1 | 1 | 0 | 4 | 1 | 5 | 1 | 22
  Male | 2 | 1 | 3 | 1 | 5 | 2 | 2 | 1 | 2 | 1 | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Adverse Event of Erythema in Part I of the Study
Description: Following topical administration of MK-0873 or matching placebo patches once daily for 21 days, the number of participants with an adverse event of erythema was recorded. An adverse event is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Time Frame: Up to Day 22 in Part 1
Population: The population consisted of all enrolled participants who received at least one dose of study medication in Part I of the study.
Measure: Number; unit: Participants
Arm/Group | Panel A - MK-0873 5.1 mg | Panel A - Placebo
Number analyzed (Participants) | 7 | 2
Participants | 0 | 0

2. Primary Outcome: Mean Maximum Plasma Concentration (Cmax) of MK-0873 Following Topical Administration for 10 Days
Description: Participant blood samples were collected on Day 11 to determine the Cmax of MK-0873 following topical administration in healthy participants and participants with psoriasis
Time Frame: Day 11
Population: The population consisted of all enrolled participants who received MK-0873 and for whom blood samples were collected and evaluable to determine Cmax.
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | Panel A - MK-0873 5.1 mg | Panel B - MK-0873 25 mg | Panel C - MK-0873 100 mg | Panel D - MK-0873 200 mg | Panel E and Extension - MK-0873 200 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
nM | NA (NA) — The value was below the lower limit of quantification. | 9.10 (1.52) | 5.22 (2.97) | 12.0 (3.41) | 9.76 (6.42)

3. Primary Outcome: Number of Participants With an Adverse Event
Description: An adverse event is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Time Frame: Up to 14 days after last dose of study drug (up to Day 42)
Population: The population consisted of all enrolled participants who received at least one dose of study medication for whom safety data were available.
Measure: Number; unit: Participants
Groups:
- Placebo - Pooled: In Parts I, II, and III, participants who received skin application of cream or patches containing placebo (and no patches containing MK-0873) were pooled for analysis.
Arm/Group | Panel A - MK-0873 5.1 mg | Panel B - MK-0873 25 mg | Panel C - MK-0873 100 mg | Panel D - MK-0873 200 mg | Panel E and Extension - MK-0873 200 mg | Placebo - Pooled
Number analyzed (Participants) | 7 | 6 | 6 | 6 | 7 | 10
Participants | 3 | 3 | 4 | 6 | 6 | 4

4. Primary Outcome: Number of Participants Who Discontinued Study Medication Due to an Adverse Event
Description: as for outcome 3
Time Frame: Up to Day 28
Population: The population consisted of all enrolled participants who received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Panel A - MK-0873 5.1 mg | Panel B - MK-0873 25 mg | Panel C - MK-0873 100 mg | Panel D - MK-0873 200 mg | Panel E and Extension - MK-0873 200 mg | Placebo - Pooled
Number analyzed (Participants) | 7 | 6 | 6 | 6 | 7 | 10
Participants | 1 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Part I: up to Day 36; Part II: up to Day 24; Part III: up to Day 42
Description: The population consisted of all enrolled participants who received at least one dose of study medication and for whom safety data were available.
Arm/Group | Panel A - MK-0873 5.1 mg | Panel B - MK-0873 25 mg | Panel C - MK-0873 100 mg | Panel D - MK-0873 200 mg | Panel E and Extension - MK-0873 200 mg | Placebo - Pooled
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6 | 0/6 | 0/6 | 0/7 | 0/10
Other Adverse Events (participants affected / at risk) | 3/7 | 3/6 | 4/6 | 6/6 | 6/7 | 4/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Panel A - MK-0873 5.1 mg (N=7) | Panel B - MK-0873 25 mg (N=6) | Panel C - MK-0873 100 mg (N=6) | Panel D - MK-0873 200 mg (N=6) | Panel E and Extension - MK-0873 200 mg (N=7) | Placebo - Pooled (N=10)
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Burning Sensation (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Headache (Nervous system disorders) | 1 | 1 | 1 | 0 | 2 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pyuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 3 | 3 | 2 | 3
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Injection-site reaction (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation.